CLINICAL TRIAL: NCT07050004
Title: Prevalence of Smoking After Lung Transplantation
Acronym: TABATRANSPLANT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00918-37
Record Dates: First submitted 2025-06-18; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Smoking; Lung Transplantation
MeSH Terms: conditions — Tobacco Smoking | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SMOKING — Patients who agree to take part in the study will complete a questionnaire covering the pre- and post-transplant aspects of smoking on their lifestyle

SUMMARY:
Smoking is one of the main risk factors for chronic obstructive pulmonary disease (COPD), the primary indication for lung transplantation (LT) in France. Resumption of smoking after transplantation is associated with an increased risk of graft dysfunction, neoplasia and reduced survival. The prevalence of resumption of smoking after transplantation is based on few data available in the literature and is estimated at between 0 and 15%. The aim of this study is to determine the prevalence of smoking in transplantation. These results will enable healthcare professionalś to carry out information, education, prevention and support actions to help patients stop smoking throughout the transplantation process.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has undergone a lung transplant (single, double or heart-lung) and is being followed up in a transplant centre in France;
* Age ≥ 18 years;
* French-speaking patient;
* Patient able to give his non-opposition.

Exclusion Criteria:

* Patient under guardianship or curatorship;
* Patient deprived of liberty ;
* Patient under court protection;
* Patients who object to the use of their data for this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have benefited from a lung or cardiopulmonary transplantation
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Assessing the prevalence of active smoking in post-lung transplantation sing a questionnaire | one year post transplantation
  Proportion of transplant patients with active smoking

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France